CLINICAL TRIAL: NCT06051422
Title: Correlation of Pelvic Asymmetry and Joint Movement During Gait in Children With Cerebral Palsy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shimaa Mohamed Reffat, Lecturer at Pediatric department of Physical therapy Faculty, Cairo University
Other Study IDs: P.T. REC/012/004462
Record Dates: First submitted 2023-07-25; First posted 2023-09-22 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Correlation of Pelvic Asymmetry and Joint Movement During Gait in Children With Cerebral Palsy
Keywords: Cerebral palsy; pelvic obliquity; joint movement
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: three dimensional formetric system — A three-dimensional computer program that automatically detects pelvic torsion, surface rotation, and anatomical landmarks. Aesculap-Meditec GMBH, based in the Netherlands, creates the Formetric Instrument System. Different subject heights could be accommodated by adjusting the scanner.
  Other Names: digital cameras

SUMMARY:
the study's particular goals were to determine whether excessive hip, knee, and ankle displacement at first contact during locomotion correlates with pelvic rotation.

ELIGIBILITY:
Inclusion Criteria:

* the lower extremities' degree of spasticity ranged from grade 1 to grade +1 on the Gross Motor Function Classification System (GMFCS) [7] classified motor function levels as being between levels I and II. Children have the cognitive ability to understand and follow instructions.

Exclusion Criteria:

* having an extensive intellectual disability, orthopedic issues, upper or lower limb surgery, visual or hearing issues, usage of behavior-altering medicines, or a major neurological illness (epilepsy)

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 20 kids with spastic cerebral palsy
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-02-12 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
pelvic asymmetry and joints movement measures | 2 months
  A three-dimensional computer program that automatically detects pelvic torsion, surface rotation, and anatomical landmarks. Aesculap-Meditec GMBH, based in the Netherlands, creates the Formetric Instrument System. Different subject heights could be accommodated by adjusting the scanner. the Unit of measures detected by degrees

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Eldoky, Egypt